CLINICAL TRIAL: NCT00642525
Title: Radiologic vs. Endoscopic Evaluation of the Conduit After Esophageal Resection: a Prospective, Blinded, Intraindividual Controlled Diagnostic Study.
Brief Title: Detection of Anastomotic Leakage After Esophageal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Jens Werner, MD Professor of Surgery, Department of Surgery, University of Heidelberg
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Endoray
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Esophageal Cancer; Anastomotic Leakage
Keywords: detection of anastomotic leakage; esophageal resection; diagnostic safety
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): A prospective, blinded, intraindividual controlled study is conducted with patients with transthoracic esophagectomy due to esophageal cancer. A radiographic contrast study is performed prior to endoscopy at the 5th to 7th postoperative day.
  Interventions: Procedure: Contrast swallow radiography, endoscopy

INTERVENTIONS:
Procedure: Contrast swallow radiography, endoscopy — Contrast swallow radiography is performed using water soluble contrast medium Esophagoscopy is performed according to standard safety guidelines

SUMMARY:
Anastomotic leakage is a major complication in esophageal surgery. Although contrast swallow is the current standard to exclude anastomotic leakage postoperatively, endoscopy may be superior. This is the first study to compare radiographic contrast study and endoscopy for the identification of local complications after subtotal esophagectomy.

DETAILED DESCRIPTION:
This prospective, blinded, intraindividual controlled study will be conducted with patients with transthoracic esophagectomy due to esophageal cancer. A radiographic contrast study will be performed prior to endoscopy at the 5th to 7th postoperative day. The investigators will not be aware of the results of the corresponding examination. Sensitivity, specificity and feasibility of the radiologic and endoscopic evaluation of the esophageal substitute will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary esophageal cancer undergoing transthoracic esophagectomy.

Exclusion Criteria:

* no transthoracic resection
* no primary anastomosis
* recurrent disease
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Detection of anastomotic leakage | 5-7 days after surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, University of Heidelberg, Heidelberg, Germany